CLINICAL TRIAL: NCT03462095
Title: Non-intensive But Non-interruptive Treatment of Adult Ph-negative Acute Lymphoblastic Leukemia With Randomization for Maintenance or Autologous Hematopoietic Stem Cell Transplantation (HSCT) Followed by Maintenance in T-cell ALL Patients
Brief Title: De-escalated Treatment Approach for Adult Ph-negative Acute Lymphoblastic Leukemia (ALL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ALL--2016
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no Auto-HSCT (No Intervention): After completing prolonged consolidation T-cell ALL patients will continue with 2 years maintenance
- Auto-HSCT (Experimental): After completing prolonged consolidation T-cell ALL patients will get autologous HSCT followed by 2 years maintenance
  Interventions: Procedure: Autologous HSCT

INTERVENTIONS:
Procedure: Autologous HSCT — After the 3rd consolidation, T-cell ALL patients, randomized to auto-HSCT will be mobilised by G-SCF and harvested disregarding MRD-status. After completing the 5th consolidation T-ALL patients will be transplanted after non-myeloablative CEAM (CCNU, Ethoposide, ARA-C, Melphalan) conditioning, and after reconstitution will continue 2-years maintenance
  Arms: Auto-HSCT

SUMMARY:
No high-dose methotrexate (MTX) and high-dose cytarabine (ARA-C) consolidation blocks, L-asparaginaseis scheduled for 1 year of treatment, 21 intrathecal injections through the whole treament, T-ALL patients in complete remossion (CR) after the informed consent are randomized to: auto-HSCT vs no auto-HSCT, - with the similar further maintenance. Stem cell harvest is performed after the 3rd consolidation by G-SCF disregarding minimal residual disease (MRD) level. Auto-HSCT is planned after the 5th consolidation phase. All primary bone samples are collected and tested for cytogenetics and molecular markers, all included patients are monitored by flow cytometry by aberrant immunophenotype in a centralized lab.

DETAILED DESCRIPTION:
* 7 days prednisolone prephase
* 8 weeks induction with de-escalation of induction chemotherapy: 3 instead of 4 dauno/vncr pulses,

  1. instead of 2 Cph injections during induction,
  2. instead of 4 ARA-C blocks, distribution of of L-asp injections through all phases
* After CR achievement T-cell ALL patients are being randomized to auto-HSCT vs no auto-HSCT
* Non-interruptive 5 consolidation phases with dose modification according to WBC and platelets count after CR achievement. Rotation of consolidation is permitted
* After the 3rd consolidation stem cells harvesting is carried out for T-cell ALL patients randomized to auto-HSCT
* Auto-HSCT after the 5th consolidation phase with non-myeloablative CEAM conditioning
* 2 years maintenance for all patients
* 21 TIT through the whole treatment with higher intensity during induction|consolidation
* Centralized MRD monitoring at +70 d, + 133 d, + 190 days; before and after auto-HSCT
* Allo-HSCT is planned only for very high risk patients (11q23 ALL, MRD positivity at day +190)

ELIGIBILITY:
Inclusion Criteria:

* age 18-55 yy, newly diagnosed non-treated Ph-negative ALL

Exclusion Criteria:

* age > 55 yy, Ph-positivity, relapsed|refractory ALL, pretreated ALL

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5-years
  Impact of autologous HSCT on DFS in T-cell ALL patients

SECONDARY OUTCOMES:
MRD-negativity after consolidation | 6 months
  Minimal Residual Disease clearance on non-intensive but non-interruptive treatment
Overall survival | 5-years
  Impact of de-escalated approach on OS

CONTACTS AND LOCATIONS:
Overall Officials: Valeriy V Savchenko, Academician, Study Director — National Research Center for hematology, Moscow, Russia
Locations (1):
- National Research Center for Hematology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Each participating site has its on-line access to WEB-data base
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once a year
Access Criteria: phone-call to coodinating center